CLINICAL TRIAL: NCT01508936
Title: A 16-Week, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Reslizumab (3.0 mg/kg) Treatment in Patients With Moderate to Severe Asthma
Brief Title: Study to Evaluate the Efficacy and Safety of Reslizumab Treatment in Patients With Moderate to Severe Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C38072/3084
Record Dates: First submitted 2012-01-03; First posted 2012-01-12 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-05

CONDITIONS: Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — reslizumab; Antibodies, Monoclonal, Humanized

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo intravenous injection every 4 weeks for a total of 4 doses.
  Interventions: Drug: Placebo
- Reslizumab 3.0 mg/kg (Experimental): Reslizumab intravenous injection at a dosage of 3.0 mg/kg every 4 weeks for a total of 4 doses.
  Interventions: Drug: Reslizumab

INTERVENTIONS:
Drug: Reslizumab — Reslizumab administered at a dosage of 3.0 mg/kg by intravenous (iv) infusion by qualified study personnel every 4 weeks for 16 weeks (for a total of 4 doses).
  Other Names: Cinquil; humanized monoclonal antibody; CEP-38072
  Arms: Reslizumab 3.0 mg/kg
Drug: Placebo — Matching placebo administered by intravenous (iv) infusion by qualified study personnel every 4 weeks for 16 weeks (for a total of 4 doses).
  Arms: Placebo

SUMMARY:
The primary objective of the study is to characterize the efficacy of reslizumab treatment, at a dosage of 3.0 milligrams per kilogram (mg/kg) every 4 weeks for a total of 4 doses, in improving pulmonary function in relation to baseline blood eosinophil levels in patients with moderate to severe asthma, as assessed by the change from baseline to week 16 in forced expiratory volume in 1 second (FEV1).

ELIGIBILITY:
Inclusion criteria:

Patients are included in the study if all of the following criteria are met:

* The patient is a man or woman, 18 through 65 years of age, with a diagnosis of asthma.
* The patient has an ACQ score of at least 1.5.
* At screening, the patient has airway reversibility of at least 12% to beta-agonist administration.
* The patient is currently taking fluticasone at a dosage of at least 440 µg daily (or equivalent). Patients' baseline asthma therapy regimens (including but not limited to inhaled corticosteroids, leukotriene antagonists, 5-lipoxygenase inhibitors, cromolyn) must be stable for 30 days before screening and continue without dosage changes throughout study.
* Female patients must be surgically sterile, 2 years postmenopausal, or must have a negative beta-human chorionic gonadotropin (ßHCG) result for a pregnancy test at screening (serum) and baseline (urine).
* Female patients of childbearing potential (not surgically sterile or 2 years postmenopausal), must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study. Acceptable methods of contraception include barrier method with spermicide, abstinence, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected).
* Written informed consent is obtained.
* The patient is in reasonable health (except for diagnosis of asthma) as judged by the investigator, and as determined by a medical history, medical examination, electrocardiogram (ECG) evaluation, serum chemistry, hematology, urinalysis, and serology.
* The patient must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period, and be willing to return to the clinic for the follow-up evaluation as specified in this protocol.

Exclusion Criteria:

Patients are excluded from participating in this study if 1 or more of the following criteria are met:

* The patient has another confounding underlying lung disorder (eg, chronic obstructive pulmonary disease, pulmonary fibrosis, lung cancer). The patient has other pulmonary conditions with symptoms of asthma and blood eosinophilia (eg, Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis).
* The patient has a clinically meaningful comorbidity that would interfere with the study schedule or procedures, or compromise the patient's safety.
* The patient has known hypereosinophilic syndrome (HES).
* The patient is a current smoker (ie, has smoked within the last 6 months prior to screening).
* The patient has a history of use of systemic immunosuppressive or immunomodulating agents (anti-immunoglobulin E [anti-IgE] mAb, methotrexate, cyclosporin, interferon-α, anti-tumor necrosis factor mAb, or omalizumab) within 6 months prior to study entry (randomization).
* The patient is currently using or has used systemic corticosteroids (includes use of oral corticosteroids) within 30 days prior to the screening visit.
* The patient is expected to be poorly compliant with study drug administration, study procedures, or visits.
* The patient has any aggravating factors that are inadequately controlled, and thus would aggravate asthma symptoms (eg, gastroesophageal reflux disease).
* The patient has participated in any investigative drug or device study within 30 days prior to screening.
* The patient has participated in any investigative biologics study within 90 days prior to screening.
* The patient has previously received reslizumab or other anti-hIL-5 mAbs (eg, mepolizumab).
* The patient is a pregnant or lactating woman. (Any women becoming pregnant during the study will be withdrawn from the study.)
* The patient has a current infection or disease that may preclude assessment of asthma.
* The patient has a history of concurrent immunodeficiency (human immunodeficiency, acquired immunodeficiency syndrome, or congenital immunodeficiency).
* The patient is suspected of current drug or alcohol abuse as specified in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria.
* The patient has presence of or suspected parasitic infestation/infection.
* Patients may not have received any live attenuated vaccine within the 12-week period before study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Respiratory Clinical Research, M.D., Study Director — Sponsor's Medical Expert
Locations (66):
- United States (66):
  - Investigational Site 861, Birmingham, Alabama
  - Investigational Site 842, Homewood, Alabama
  - Investigational Site 887, Jasper, Alabama
  - Investigational Site 809, Tucson, Arizona
  - Investigational Site 892, Tucson, Arizona
  - Investigational Site 846, Little Rock, Arkansas
  - Investigational Site 828, Anaheim, California
  - Investigational Site 900, Fresno, California
  - Investigational Site 862, Huntington Beach, California
  - Investigational Site 852, Los Angeles, California
  - Investigational Site 909, Los Angeles, California
  - Investigational Site 864, Newport Beach, California
  - Investigational Site 812, Rancho Mirage, California
  - Investigational Site 808, Riverside, California
  - Investigational Site 804, Sacramento, California
  - Investigational Site 837, Centennial, Colorado
  - Investigational Site 851, Denver, Colorado
  - Investigational Site 832, Wheat Ridge, Colorado
  - Investigational Site 855, Jacksonville, Florida
  - Investigational Site 865, Miami, Florida
  - Investigational Site 881, Miami, Florida
  - Investigational Site 805, Albany, Georgia
  - Investigational Site 870, Stockbridge, Georgia
  - Investigational Site 816, Chicago, Illinois
  - Investigational Site 824, Shiloh, Illinois
  - Investigational Site 883, Evansville, Indiana
  - Investigational Site 878, Fort Wayne, Indiana
  - Investigational Site 820, Lenexa, Kansas
  - Investigational Site 873, Owensboro, Kentucky
  - Investigational Site 801, Lafayette, Louisiana
  - Investigational Site 877, Mandeville, Louisiana
  - Investigational Site 875, White Marsh, Maryland
  - Investigational Site 871, Fall River, Massachusetts
  - Investigational Site 834, North Dartmouth, Massachusetts
  - Investigational Site 889, Troy, Michigan
  - Investigational Site 838, Rolla, Missouri
  - Investigational Site 818, St Louis, Missouri
  - Investigational Site 841, St Louis, Missouri
  - Investigational Site 857, Albuquerque, New Mexico
  - Investigational Site 819, Newburgh, New York
  - Investigational Site 844, Charlotte, North Carolina
  - Investigational Site 845, Middleburg Heights, Ohio
  - Investigational Site 810, Tulsa, Oklahoma
  - Investigational Site 859, Ashland, Oregon
  - Investigational Site 859, Portland, Oregon
  - Investigational Site 854, Jenkintown, Pennsylvania
  - Investigational Site 843, Providence, Rhode Island
  - Investigational Site 802, Florence, South Carolina
  - Investigational Site 814, Orangeburg, South Carolina
  - Investigational Site 821, Spartanburg, South Carolina
  - Investigational Site 829, Spartanburg, South Carolina
  - Investigational Site 850, Knoxville, Tennessee
  - Investigational Site 803, Nashville, Tennessee
  - Investigational Site 880, Dallas, Texas
  - Investigational Site 858, Dickinson, Texas
  - Investigational Site 869, Live Oak, Texas
  - Investigational Site 879, Plano, Texas
  - Investigational Site 847, Salt Lake City, Utah
  - Investigational Site 876, West Jordan, Utah
  - Investigational Site 840, Fairfax, Virginia
  - Investigational Site 836, Richmond, Virginia
  - Investigational Site 867, Seattle, Washington
  - Investigational Site 833, Spokane, Washington
  - Investigational Site 904, Vancouver, Washington
  - Investigational Site 806, Greenfield, Wisconsin
  - Investigational Site 823, La Crosse, Wisconsin

REFERENCES:
- [Derived] Corren J, Weinstein S, Janka L, Zangrilli J, Garin M. Phase 3 Study of Reslizumab in Patients With Poorly Controlled Asthma: Effects Across a Broad Range of Eosinophil Counts. Chest. 2016 Oct;150(4):799-810. doi: 10.1016/j.chest.2016.03.018. Epub 2016 Mar 25. PMID 27018175

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 869 patients were screened for enrollment into this study. Of the 869 patients screened, 511 patients at 103 centers in the US met entry criteria and were considered to be eligible for enrollment into the study.
Pre-assignment Details: Randomization was stratified by occurrence of asthma exacerbation(s) during the previous year (yes or no). Within each stratum, patients were randomly assigned in a 4:1 ratio to receive treatment with reslizumab at 3.0 mg/kg or matching placebo.
Period: Overall Study
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Started | 102 | 409
Randomized, Not Analyzed | 4 (Participants from two centers were omitted from all analyses.) | 11 (Participants from two centers were omitted from all analyses.)
Randomized | 98 | 398
Randomized, Not Treated | 1 | 3
Safety Analysis Set | 97 | 395
Full Analysis Set | 97 | 395
FEV1 Subpopulation Analysis Set | 91 | 346
Completed | 79 | 330
Not Completed | 23 | 79
Not completed — Adverse Event | 11 | 32
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 4 | 18
Not completed — Protocol Violation | 2 | 3
Not completed — Lost to Follow-up | 2 | 9
Not completed — Other | 0 | 5
Not completed — Data from 2 sites deemed invalid | 4 | 11

BASELINE CHARACTERISTICS:
Population: Randomized, analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Reslizumab 3.0 mg/kg | Total
Number analyzed (Participants) | 98 | 398 | 496
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (13.38) | 44.9 (12.00) | 44.9 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 261 | 315
  Male | 44 | 137 | 181
Race/Ethnicity, Customized [Number; unit: participants]
  White | 73 | 260 | 333
  Black | 21 | 113 | 134
  Asian | 2 | 10 | 12
  American Indian or Alaskan Native | 0 | 3 | 3
  Pacific Islander | 2 | 0 | 2
  Other | 0 | 12 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic and Non-Latino | 90 | 354 | 444
  Hispanic or Latino | 8 | 44 | 52
Weight [Mean (Standard Deviation); unit: kg] | 90.9 (20.68) | 90.6 (23.92) | 90.7 (23.30)
Height [Mean (Standard Deviation); unit: cm] | 169.7 (10.25) | 167.7 (10.35) | 168.1 (10.35)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (6.66) | 32.2 (8.69) | 32.2 (8.33)
Asthma Control Questionnaire (ACQ) [Mean (Standard Deviation); unit: units on a scale] — n=98, 396, 494 The ACQ score was measured using the ACQ-7. Six questions are-self assessments; the seventh item is the result of the patient's % predicted FEV1 measurement. Each item has 7 possible answers on a scale of 0 to 6, and the total score is the mean of all responses (the total scale is therefore 0-6). A score of 0 indicates good asthma control; higher scores indicate increasingly poorer asthma control.
  units on a scale | 2.564 (0.6909) | 2.558 (0.6992) | 2.559 (0.6969)
Forced Expiratory Volume in 1 second (FEV1) [Mean (Standard Deviation); unit: liters] — n=98, 396, 494
  liters | 2.180 (0.6355) | 2.101 (0.6950) | 2.117 (0.6837)
Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: liters] — n=98, 396, 494
  liters | 3.215 (0.9076) | 3.047 (0.9577) | 3.081 (0.9494)
Forced Expiratory Flow at 25% to 75% of the Forced Vital Capacity (FEF25%-75%) [Mean (Standard Deviation); unit: liters/second] — n=96, 393, 489
  liters/second | 1.553 (0.6791) | 1.650 (0.9037) | 1.631 (0.8645)
Percent Predicted Forced Expiratory Volume in 1 Second (% predicted FEV1) [Mean (Standard Deviation); unit: % predicted] — n=98, 396, 494
  % predicted | 66.5 (15.53) | 66.8 (16.26) | 66.7 (16.10)
Blood Eosinophil Counts [Mean (Standard Deviation); unit: 10^9 blood eosinophil/liter] — n=96, 397, 493
  10^9 blood eosinophil/liter | 0.277 (0.2209) | 0.281 (0.2448) | 0.280 (0.2401)
Average Daily Use of Short-Acting Beta-Agonist Therapy (SABA) in Past 3 Days [Mean (Standard Deviation); unit: puffs of SABA/day] — n=98, 395, 493
  puffs of SABA/day | 2.0 (1.82) | 1.9 (1.84) | 1.9 (1.83)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 16 in Full Analysis Set
Description: FEV1 is a standard measurement of air movement in the lungs of patients with asthma. It is the volume of air expired in the first second of a forced expiration. Improvement in FEV1 is a measure in the reduction of bronchospasm, the reduction of airway inflammation, or both. FEV1 was measured using forced expiratory air spirometry.
  Data represent the slope estimate of change from baseline in FEV1 (measured in liters) at Week 16 versus baseline eosinophil count (measured in 10^9/liter) by treatment group.
Time Frame: Baseline (Day 1), Week 16
Population: Full analysis set (FAS) includes randomized patients treated with at least 1 dose of study drug, and had assessments in the timeframes. Pulmonary function tests were excluded if a limited subset of medications that could significantly confound interpretation were used within 7 days of scheduled visits.
Measure: Mean (Standard Error); unit: FEV1 liters/ eosinophils 10^9/liter
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 83 | 344
FEV1 liters/ eosinophils 10^9/liter | -0.2778 (0.2379) | 0.0229 (0.0944)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; The primary analysis was the linear regression model with model effects including treatment (reslizumab or placebo), blood eosinophil count at baseline, and the interaction of treatment and eosinophil count. A significant treatment by baseline eosinophil interaction would indicate that treatment difference varies by the baseline eosinophil count; Test type: Superiority or Other; p = 0.2407, Regression, Linear — The interaction was tested at the significance level 0.10 using the FAS; slope difference = 0.3007, Standard Error of Mean 0.2559 — Active - Placebo

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Over 16 Weeks Using Mixed Model for Repeated Measures
Description: FEV1 is a standard measurement of air movement in the lungs of patients with asthma. It is the volume of air expired in the first second of a forced expiration. Improvement in FEV1 is a measure in the reduction of bronchospasm, the reduction of airway inflammation, or both. FEV1 was measured using forced expiratory air spirometry. Positive change from baseline scores indicate improvement in asthma control.
  During study (Weeks 4, 8, 12 and 16) average value was calculated using a mixed effects model for repeated measures (MMRM) with treatment (reslizumab or placebo), blood eosinophil count at baseline, and the interaction of treatment and eosinophil count as a random effect.
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16
Population: Full analysis set (FAS) includes randomized patients treated with at least 1 dose of study drug, and contributed at least once to the analysis. Pulmonary function tests were excluded if a limited subset of medications that could significantly confound interpretation were used within 7 days of scheduled visits.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 96 | 390
liters | 0.175 (0.0377) | 0.251 (0.0200)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; The change from baseline over the 16 week treatment period was measured for the key secondary variables of: * Lung function as measured by FEV1 * ACQ Testing of the key secondary variables was performed using the sequential testing procedure in the order as specified above at the alpha level of 0.05; Test type: Superiority or Other; p = 0.0697, Regression, Linear — Statistical significance level is 0.05; treatment, blood eosinophil count at baseline, and the interaction of treatment and eosinophil count as fixed effects; Mean Difference (Final Values) = 0.076, 95% CI 2-sided [-0.006 to 0.158], Standard Error of Mean 0.0417 — Active - Placebo

3. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) Over 16 Weeks Using Mixed Model for Repeated Measures
Description: The ACQ score was measured using the ACQ-7. Six questions are-self assessments; the seventh item is the result of the patient's % predicted FEV1 measurement. Each item has 7 possible answers on a scale of 0 to 6, and the total score is the mean of all responses (the total scale is therefore 0-6). A score of 0 indicates good asthma control; higher scores indicate increasingly poorer asthma control. Negative change from baseline scores indicate improvement in asthma control.
  During study (Weeks 4, 8, 12 and 16) average value was calculated from mixed model repeated measures (MMRM) with treatment, visit, treatment by visit interaction, history of asthma exacerbation in the previous year, height, baseline value, and sex as fixed factors, and patient as a random effect.
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16
Population: Full analysis set of participants who contributed at least once to the analysis. ACQ were excluded from the FAS if they were obtained at scheduled visits which were preceded by usage within 7 days of a limited subset of medications that could significantly confound interpretation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 96 | 390
units on a scale | -0.614 (0.0689) | -0.737 (0.0364)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1072, t-test, 2 sided — significance level of 0.05; Fixed effects for treatment, hx of asthma exacerbation, sex, visit, and interaction of treatment and visit; covariates for height and baseline value; Mean Difference (Final Values) = -0.123, 95% CI 2-sided [-0.273 to 0.027], Standard Error of Mean 0.0762 — Active - Placebo

4. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 16 in FEV1 Subpopulation
Description: FEV1 is a standard measurement of air movement in the lungs of patients with asthma. It is the volume of air expired in the first second of a forced expiration. Improvement in FEV1 is a measure in the reduction of bronchospasm, the reduction of airway inflammation, or both. FEV1 was measured using forced expiratory air spirometry.
  As with the primary outcome, data represent the slope estimate of change from baseline in FEV1 (measured in liters) at Week 16 versus baseline eosinophil count (measured in 10^9/liter) by treatment group. However the FEV1 subpopulation includes participants with more impaired lung function (% predicted FEV1 <85% at baseline).
Time Frame: Baseline (Day 1), Week 16
Population: The FEV1 sub-population analysis set includes all participants in the FAS with % predicted FEV1 <85% at baseline. Pulmonary function tests were excluded if a limited subset of medications that could significantly confound interpretation were used within 7 days of scheduled visits.
Measure: Mean (Standard Error); unit: FEV1 liters/ eosinophils 10^9/liter
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 91 | 346
FEV1 liters/ eosinophils 10^9/liter | -0.2944 (0.2443) | 0.0271 (0.1019)

5. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Weeks 4, 8, 12, and 16
Description: FEV1 is a standard measurement of air movement in the lungs of patients with asthma. It is the volume of air expired in the first second of a forced expiration. Improvement in FEV1 is a measure in the reduction of bronchospasm, the reduction of airway inflammation, or both. FEV1 was measured using forced expiratory air spirometry. Positive change from baseline scores indicate improvement in asthma control.
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, and 16
Population: Full analysis set. Number of participants analyzed represents # with FEV1 baseline values (one reslizumab participant was missing a valid baseline FEV1.) Number participants with assessments in the timeframes are listed with the time designation.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 97 | 394
liters
  Week 4 (n= 96, 386) | 0.164 (0.0395) | 0.224 (0.0208)
  Week 8 (n= 93, 377) | 0.199 (0.0421) | 0.249 (0.0220)
  Week 12 (n= 90, 357) | 0.152 (0.0430) | 0.277 (0.0226)
  Week 16 (n=83, 344) | 0.187 (0.0446) | 0.255 (0.0232)

6. Secondary Outcome: Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (% Predicted FEV1) at Weeks 4, 8, 12, 16 and Endpoint
Description: The percent predicted FEV1 is the ratio of the volume of air expired in the first second of a forced expiration to the patient's predicted FEV based on a similar population without asthma. Percent predicted lung function values were transcribed directly from the lung function report to the CRF, without any calculation by Teva. Positive change from baseline scores indicate improvement in asthma control.
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, and 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 97 | 394
percentage of predicted FEV1
  Week 4 (n=96, 385) | 4.8 (9.83) | 6.7 (12.26)
  Week 8 (n=93, 377) | 6.0 (9.9) | 7.2 (13.41)
  Week 12 (n=90, 357) | 4.2 (10.36) | 8.2 (13.23)
  Week 16 (n=83, 344) | 5.5 (11.76) | 7.8 (13.60)
  Endpoint (n=96, 390) | 5.2 (11.76) | 7.5 (13.26)

7. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Weeks 4, 8, 12, and 16
Description: The FVC is the volume of air that can be forcibly blown out after full inspiration, measured in liters. FV was measured using forced expiratory air spirometry. Positive change from baseline scores indicate improvement in asthma control.
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, and 16
Population: Full analysis set. Number of participants analyzed represents # with FVC baseline values (one reslizumab participant was missing a valid baseline FVC.) Number participants with assessments in the timeframes are listed with the time designation.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 97 | 394
liters
  Week 4 (n=96, 386) | 0.167 (0.0469) | 0.235 (0.0247)
  Week 8 (n=93, 377) | 0.179 (0.0474) | 0.243 (0.0249)
  Week 12 (n=90, 357) | 0.176 (0.0500) | 0.284 (0.0263)
  Week 16 (n=84, 345) | 0.234 (0.0506) | 0.246 (0.0264)

8. Secondary Outcome: Change From Baseline in the Forced Expiratory Flow at 25% to 75% of the Forced Vital Capacity (FEF25%-75%) at Weeks 4, 8, 12, and 16
Description: The FEF25%-75% is the forced expiratory flow at 25% to 75% of the forced vital capacity. FEF25%-75% was measured using forced expiratory air spirometry. Positive change from baseline scores indicate improvement in asthma control.
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, and 16
Population: Full analysis set. Number of participants analyzed represents # with FEF25%-75% baseline values. Number of participants with assessments in the timeframes are listed with the time designation.
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 95 | 391
liters/second
  Week 4 (n=93, 382) | 0.210 (0.0565) | 0.184 (0.0295)
  Week 8 (n=90, 374) | 0.270 (0.0609) | 0.240 (0.0315)
  Week 12 (n=87, 354) | 0.136 (0.0635) | 0.256 (0.0329)
  Week 16 (n=82, 342) | 0.179 (0.0875) | 0.241 (0.0441)

9. Secondary Outcome: Change From Baseline in Average Daily Use of Short-Acting Beta-Agonist Therapy (SABA) at Weeks 4, 8, 12, and 16
Description: SABA are used for quick relief of asthma symptoms. The number of times SABA therapy was used was assessed using 3 day recall at scheduled visits. Participants were asked to recall whether SABAs were used within 3 days of the scheduled visit and, if so, how many puffs were used. Daily use was the average of those 3 days. Negative change from baseline scores indicate improvement in asthma control.
Time Frame: Baseline (Day -2 to 1), Weeks 4, 8, 12, and 16
Population: Full analysis set. Number of participants analyzed represents # with SABA use baseline values. Number participants with assessments in the timeframes are listed with the time designation.
Measure: Least Squares Mean (Standard Error); unit: puffs of SABA/day
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 96 | 392
puffs of SABA/day
  Week 4 (n=96, 388) | -0.1 (0.19) | -0.2 (0.10)
  Week 8 (n=94, 377) | -0.2 (0.18) | -0.3 (0.09)
  Week 12 (n=89, 356) | -0.2 (0.20) | -0.3 (0.10)
  Week 16 (n=84, 345) | -0.4 (0.18) | -0.3 (0.09)

10. Secondary Outcome: Change From Baseline in Blood Eosinophil Counts at Weeks 4, 8, 12, 16, Follow-up (Week 28) and Endpoint
Description: Blood eosinophil counts were measured using a standard complete blood count with differential blood test at each scheduled visit. Follow-up was performed approximately 12 weeks after the 16 week treatment period. Endpoint is the last post-baseline assessment.
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16, Follow-up (Week 28)
Population: Full analysis set. Number of participants analyzed represents # with blood eosinophil count baseline values. Number participants with assessments in the timeframes are listed with the time designation.
Measure: Mean (Standard Deviation); unit: 10^9/liter
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 95 | 394
10^9/liter
  Week 4 (n=93, 385) | 0.010 (0.1917) | -0.226 (0.2297)
  Week 8 (n=91, 372) | 0.036 (0.3104) | -0.239 (0.2389)
  Week 12 (n=84, 353) | 0.027 (0.2082) | -0.240 (0.2418)
  Week 16 (n=80, 346) | 0.021 (02466) | -0.239 (0.2462)
  Follow-up (n=90, 364) | 0.035 (0.3369) | -0.159 (0.2301)
  Endpoint (n=94, 392) | 0.036 (0.3306) | -0.169 (0.2294)

11. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) at Weeks 4, 8, 12 and 16
Description: The ACQ score was measured using the ACQ-7. Six questions are self-assessments; the seventh item is the result of the patient's % predicted FEV1 measurement. Each item has 7 possible answers on a scale of 0 to 6, and the total score is the mean of all responses (the total scale is therefore 0-6). A score of 0 indicates good asthma control; higher scores indicate increasingly poorer asthma control. Negative change from baseline scores indicate improvement in asthma control.
Time Frame: Baseline (Day 1), Weeks 4, 8, 12 and 16
Population: Full analysis set. Number of participants analyzed represents # with ACQ baseline values. Number participants with assessments in the timeframes are listed with the time designation. ACQ were excluded if obtained at visits which were preceded by usage within 7 days of a limited subset of medications that could significantly alter interpretation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 97 | 394
units on a scale
  Week 4 (n=96, 385) | -0.502 (0.0710) | -0.585 (0.0375)
  Week 8 (n=93, 377) | -0.631 (0.0807) | -0.701 (0.0420)
  Week 12 (n=90, 357) | -0.674 (0.0843) | -0.818 (0.0439)
  Week 16 (n=83, 343) | -0.648 (0.0878) | -0.844 (0.0453)

12. Secondary Outcome: Participants With Treatment-Emergent Adverse Events
Description: An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an inability to carry out usual activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Week 28
Population: The safety analysis set includes all patients who took at least 1 dose of study drug, regardless of whether the patients were randomized.
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 97 | 395
participants
  Any adverse event | 72 | 218
  Severe adverse event | 10 | 25
  Treatment-related adverse event | 16 | 28
  Deaths | 0 | 0
  Serious AEs other than death | 4 | 16
  Treatment-related serious AE | 0 | 2
  Withdrawn from study due to adverse events | 12 | 29
  Withdrawn from study due to treatment-related AE | 1 | 3

13. Secondary Outcome: Participants With Treatment-Emergent Potentially Clinically Significant (PCS) Abnormal Lab Values
Description: Data represents participants with potentially clinically significant (PCS) abnormal serum chemistry, hematology, and urinalysis values during any of the lab tests conducted during the treatment period.
  Significance criteria:
  * Blood urea nitrogen: >=10.71 mmol/L
  * Creatinine: >=177 μmol/L
  * Uric acid: M>=625, F>=506 μmol/L
  * Aspartate aminotransferase: >=3*upper limit of normal (ULN). Normal range is 10-43 U/L
  * Alanine aminotransferase: >=3*ULN. Normal range is 10-40 U/L
  * GGT = gamma-glutamyl transpeptidase: >= 3*ULN. Normal range is 4-49 U/L.
  * Total bilirubin: >=34.2 μmol/L
  * Creatinine phosphokinase: >5*ULN. Normal range is 24-207 U/L.
  * White blood cells: <=3.0 or >20 10^9/L
  * Hemoglobin: M<=115, F<=95 g/dL
  * Hematocrit: M<0.37, F<0.32 L/L
  * Platelets: <=75 10^9/L
  * Absolute neutrophil count: <=1.0 10^9/L
  * Urinalysis: blood, glucose, ketones and total protein: >=2 unit increase from baseline
Time Frame: Week 4 to Week 16
Population: Safety analysis set with assessments
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 97 | 393
participants
  Atleast 1 PCS abnormal serum blood chemistry value | 8 | 26
  Blood urea nitrogen | 0 | 7
  Creatinine | 0 | 1
  Uric acid | 1 | 7
  Aspartate aminotransferase | 1 | 3
  Alanine aminotransferase | 3 | 5
  GGT | 2 | 11
  Total bilirubin | 1 | 0
  Creatinine phosphokinase | 1 | 11
  At least 1 PCS abnormal hematology value | 4 | 30
  White blood cells - low | 0 | 6
  White blood cells - high | 0 | 4
  Hemoglobin | 0 | 10
  Hematocrit | 1 | 19
  Platelets | 0 | 1
  Absolute neutrophil count | 3 | 7
  At least 1 PCS abnormal urinalysis value | 23 | 94
  Blood (hemoglobin) | 6 | 40
  Glucose | 3 | 17
  Ketones | 6 | 7
  Total protein | 11 | 43

14. Secondary Outcome: Participants With Treatment-Emergent Potentially Clinically Significant (PCS) Vital Signs Values
Description: Data represents participants with potentially clinically significant (PCS) vital sign values during any of the treatment period exams.
  Significance criteria
  * Heart rate - high: >100 and increase of >= 30 beats/minute (bpm)
  * Sitting systolic blood pressure - high: >160 and increase of >=30 mmHg
  * Sitting systolic blood pressure - low: <90 and decrease of >=30 mmHg
  * Sitting diastolic blood pressure - high: >100 and increase of >=12 mmHg
  * Sitting diastolic blood pressure - low: <50 and decrease of >=12 mmHg
  * Body temperature - high: >100.5° Fahrenheit or 38.1° Celsius and increase of >2°
  * Body temperature - low: <96.5° Fahrenheit or <35.8° Celsius
Time Frame: Week 4 to Week 28
Population: Safety analysis set of participants with assessments
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 97 | 394
participants
  At least 1 PCS abnormality | 7 | 43
  Heart rate | 0 | 4
  Sitting systolic blood pressure - high | 1 | 6
  Sitting systolic blood pressure - low | 1 | 4
  Sitting diastolic blood pressure - high | 2 | 3
  Sitting diastolic blood pressure - low | 0 | 2
  Body temperature - high | 1 | 2
  Body temperature - low | 2 | 25

15. Secondary Outcome: Participants With Treatment-Emergent Potentially Clinically Significant (PCS) Electrocardiogram (ECG) Abnormalities
Description: Counts represent the number of participants with potentially clinically significant ECG abnormalities as assessed by the investigator.
Time Frame: Week 16 or endpoint
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 97 | 395
participants | 0 | 1

16. Secondary Outcome: Participants With a Positive Anti-Reslizumab Antibody Status During Study
Description: Counts of participants with a positive anti-drug antibody (ADA) response during treatment is offered for the experimental treatment arm. Blood samples were collected for determination of ADAs before study drug infusion at screening, weeks 8 and 16 or early withdrawal. Serum samples from patients who were treated with reslizumab were analyzed for ADA by Teva (Teva Biopharmaceuticals USA, Rockville, MD) using a validated homogeneous solution-based bridging enzyme-linked immunosorbent assay (ELISA).
  Endpoint =week 16 or early withdrawal.
  Counts represent the total number of participants at each time point with a positive immunogenicity test, and not 'new' participants with a positive test. An overall status of positive includes participants who had a positive ADA at any time point.
Time Frame: Screening (Week -3), Weeks 8 and 16
Population: Safety analysis set; antibody assessments reported for active treatment arm only.
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 0 | 395
participants
  Overall status - negative |  | 376
  Overall status - positive |  | 19
  Screening status - negative |  | 375
  Screening status - positive |  | 13
  Week 8 - negative |  | 346
  Week 8 - positive |  | 15
  Week 16 - negative |  | 328
  Week 16 - positive |  | 9
  Endpoint - negative |  | 375
  Endpoint - positive |  | 10

ADVERSE EVENTS:
Time Frame: Day 1 to Week 28
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 4/97 | 16/395
Other Adverse Events (participants affected / at risk) | 41/97 | 118/395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=97) | Reslizumab 3.0 mg/kg (N=395)
Neurogenic bowel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral vasoconstriction (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=97) | Reslizumab 3.0 mg/kg (N=395)
Nausea (Gastrointestinal disorders) | 5 (6) | 3 (3)
Bronchitis (Infections and infestations) | 6 (7) | 14 (14)
Nasopharyngitis (Infections and infestations) | 5 (5) | 13 (15)
Sinusitis (Infections and infestations) | 7 (7) | 22 (26)
Upper respiratory tract infection (Infections and infestations) | 11 (13) | 42 (50)
Asthma (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 48 (58)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.